CLINICAL TRIAL: NCT04172090
Title: Short-term Effects of Physical Inactivity on Insulin Sensitivity, Appetite, Energy Balance, and Cardiovascular Responses in Healthy Humans.
Brief Title: Effects of Physical Inactivity on Insulin Sensitivity, Appetite, Energy Balance, and Cardiovascular Responses in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: I200317
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2019-11

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): 2 consecutive days of standardised daily levels of moderate physical activity (PAL=1.85 reflecting their habitual levels), and matched energy (food) intake
  Interventions: Other: Control
- SIT+E (Experimental): 2 consecutive days of reduced physical activity induced by prolonged periods of sitting (PAL=1.4) whilst maintaining the level of food intake prescribed in the Control trial, thus creating a positive energy balance
  Interventions: Other: SIT+E
- SIT=E (Experimental): 2 consecutive days of reduced physical activity induced by prolonged periods of sitting (PAL=1.4) whilst reducing food intake to match the reduction in energy expenditure induced by inactivity, thus maintaining energy balance
  Interventions: Other: SIT=E

INTERVENTIONS:
Other: Control — Normal physical activity and standard energy intake
  Arms: Control
Other: SIT+E — Reduced physical activity and standard energy intake
  Arms: SIT+E
Other: SIT=E — Reduced physical activity and reduced energy intake
  Arms: SIT=E

SUMMARY:
Physical inactivity is a significant predictor of major non-communicable diseases such as type 2 diabetes (7%), cardiovascular disease (6%), musculoskeletal disorders and some cancers, and has been proposed to be the 4th leading cause of death worldwide. Reduced physical activity leads to an impaired function of the hormone insulin and increased adiposity. Thus, the elimination of physical inactivity would remove between 6% and 10% of the major non-communicable diseases and increase life expectancy. The aim of the study is to investigate the effects of a short-term (2-day) period of reduced physical activity, with and without a proportional decrease in energy intake, on the action of insulin to regulate blood sugar fluctuations, appetite, and cardiovascular parameters (heart rate, cardiac output, stroke volume, blood flow, arterial blood pressure, peripheral vascular resistance) in response to food ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Males and females
* Age (18-35 years old)
* Body mass index (BMI) of 18-27 kg/m2
* Waist circumference <94cm for males and <80cm for females
* Ability to give informed consent

Exclusion Criteria:

* Smoking
* Any metabolic (e.g. diabetes), endocrine (e.g. hyperthyroidism) or cardiovascular (e.g. heart or blood) abnormalities including hypertension or heart failure
* Clinically significant abnormalities on screening including ECG abnormalities
* Taking routine medication that may alter cardiovascular function and blood flow (e.g. blood pressure-lowering drugs or drugs that cause hypertension)
* Well trained individuals with PAL>2.00; on an energy-restricted diet or seeking to lose weight
* High alcohol consumption (<3-4 units/d for men; <2-3 units/d for women)
* Females who are pregnant or lactating; self-reported allergy, intolerance or strong dislike of foods or drinks to be offered for the test breakfast, pasta meal or during the intervention period
* Beck Depression Inventory score >10 and Eating Attitudes Test (EAT-26) score >20 as self-reported markers of symptoms and concerns characteristic of depression and eating disorders, respectively.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
The incremental area under curve for Insulin | Over three hours from baseline
  The incremental area under curve for Insulin will be calculated using samples collected at 20 minute intervals between baseline and three hours

SECONDARY OUTCOMES:
The incremental area under curve for arterialized whole blood glucose | Over four hours from baseline
  The incremental area under curve for arterialized whole blood glucose will be calculated using samples collected at 10 minute intervals between baseline and four hours

OTHER OUTCOMES:
The incremental area under curve for free fatty acids | Over three hours from baseline
  The incremental area under curve for free fatty acids will be calculated using samples collected at 20 minute intervals between baseline and three hours
The incremental area under curve for Triglycerides | Over three hours from baseline
  The incremental area under curve for Triglycerides will be calculated using samples collected at 20 minute intervals between baseline and three hours
The incremental area under curve for Ghrelin | Over four hours from baseline
  The incremental area under curve for Ghrelin will be calculated using samples collected at one hour intervals between baseline and four hours
The incremental area under curve for composite satiety score | Over four hours from baseline
  Composite satiety score will be calculated using 100mm visual analogue score ratings of satiety, fullness, hunger, desire to eat and prospective food consumption collected every 20 minutes between baseline and four hours.
Weight of consumption of a pasta meal three hours after baseline | Three hours post baseline
  Weight of pasta consumed from a bowel refilled prior to being empty until participants feel comfortably full
The incremental area under curve for cardiovascular parameters | Over three hours from baseline
  The incremental area under curve for mean blood pressure,cardiac output, stroke volume, peripheral resistance, heart rate, systolic blood pressure and diastolic blood pressure continuously over three hours from baseline using Finometer
The incremental area under curve for limb blood flow | Over three hours from baseline
  The incremental area under curve for limb blood flow measured at 30 minute intervals between baseline and three hours using venous occlusion plethysmography

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
only anonymised individual personal data will be shared, upon specific request from other researchers, for example, in order to undertake a meta analysis